CLINICAL TRIAL: NCT06965738
Title: Buccal Fat Applied to Transoral Robotic Lateral Oropharyngectomy Defects to Lessen Radical Tonsillectomy Pain (BOLT)
Brief Title: Buccal Fat for Transoral Robotic Lateral Oropharyngectomy Defects to and Postoperative Pain
Acronym: BOLT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Christopher Yao, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-5894
Record Dates: First submitted 2025-03-31; First posted 2025-05-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Tonsil Neoplasm; Oropharynx Neoplasm; Transoral Robotic Surgery
Keywords: Transoral Robotic Surgery; Buccal Fat; Postoperative Pain
MeSH Terms: conditions — Tonsillar Neoplasms; Oropharyngeal Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transoral lateral oropharyngectomy alone (Active Comparator): Transoral lateral oropharyngectomy without buccal fat reconstruction
  Interventions: Procedure: No buccal fat reconstruction
- Transoral lateral oropharyngectomy with buccal fat reconstruction (Experimental): Transoral lateral oropharyngectomy with buccal fat reconstruction
  Interventions: Procedure: Buccal fat reconstruction

INTERVENTIONS:
Procedure: Buccal fat reconstruction — Ipsilateral buccal fat rotation flap for reconstruction of lateral oropharyngectomy defect
  Arms: Transoral lateral oropharyngectomy with buccal fat reconstruction
Procedure: No buccal fat reconstruction — No reconstruction of lateral oropharyngectomy defect
  Arms: Transoral lateral oropharyngectomy alone

SUMMARY:
The goal of this randomized clinical trial is to determine the pain intensity during rest and swallowing in patients undergoing transoral robotic surgery for tonsil lesions with and without buccal fat reconstruction. The main question it aims to answer is: does buccal fat after transoral robotic surgery reduce pain after surgery? Additional questions to be explored include if there is a difference in swallowing, complication rates, pain medication usage, and feeding tube usage. Participants will be asked to rate their pain and swallowing on a visual analogue scale after surgery. The group will be compared compared to a control group that undergoes transoral robotic surgery without buccal fat reconstruction.

DETAILED DESCRIPTION:
Trans-oral robotic surgery (TORS) for oropharyngeal cancers have transformed how oropharyngeal cancers are managed, allowing for minimally invasive surgical access to remove tumors of the tonsil and base of tongue. While large incisions and open approaches can be avoided, oropharyngeal defects following TORS are traditionally left as an open wound to heal by secondary intention, resulting in significant postoperative pain, and possibly dysphagia and dehydration.

While this has been highlighted as a key outcome measure, studies on acute pain following TORS have not had any standardization regarding the timing of pain measurement, and pain assessment. Only one study has assessed pain during 'movement-related pain', such as swallowing, which has been advocated as a key metric. Most studies used a visual analogue scale, however, majority failed to describe the timing of pain assessment relative to administration of analgesia, time of day, or diet. Overall, pain ratings and opioid utilization were highly variable between studies resulting in pain ratings ranging widely from 2.5-8 in the first few days postoperatively.

Based on the current evidence, multimodal analgesia resulted in the lowest pain ratings following TORS, with those that included gabapentin, a COX-2 inhibitor and acetaminophen having excellent pain control in the early postoperative period. Using these regimens, Castellanos et al. found that postoperative opioid consumption significantly decreased in the first three postoperative days. Clayburgh, et al. identified that addition of perioperative corticosteroids was safe and significantly improved diet consistency, and decreased length of hospital stay, though pain scores were minimally affected.

No study thus far has assessed the impact of surgical interventions on postoperative pain and swallowing. This single center, phase II, randomized control trial aims to evaluate the impact of the buccal fat rotational flap on the postoperative pain following TORS.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Require a transoral robotic lateral oropharyngectomy as a result of the following conditions :

   * Early - intermediate stage tonsillar squamous cell carcinoma (T1-2N0-1 p16+/- SCC of the palatine tonsils)
   * Early -intermediate stage salivary gland tumors of the palatine tonsils
   * based on FNA, Core biopsy, Punch biopsy
3. Ability to understand and willing to sign a written informed consent

Exclusion Criteria:

1. History of prior head and neck squamous cell carcinoma, or prior head and neck radiotherapy
2. Presence of retropharyngeal lymphadenopathy
3. Presence of bilateral lymphadenopathy, or patients requiring bilateral neck dissections.
4. Patients with trismus at baseline
5. Patients with psychological risk factors for persistent opioid use or drug addiction
6. Need for open surgery (transcervical lateral oropharyngectomy), free tissue transfer, or alternative regional flap.
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain during rest and swallowing | Once each at the following timepoints: 1-2 week preoperatively, postoperative day 1-3, postoperative day 7-10, postoperative day 21-28
  Postoperative pain during rest and swallowing on visual analogue scale at multiple time points

SECONDARY OUTCOMES:
Surgical Complications | 30 days postoperatively
  Surgical complications and adverse events within 30 days postoperatively using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC-AE v4.0)
Opioid usage | 30 days postoperatively
  Determine opioid usage
Postoperative Hemorrhage | 30 days postoperatively
  Postoperative hemorrhage after TORS
Speech and Swallowing | Once each at the following timepoints: 1-2 week preoperatively, postoperative day 7-10, postoperative day 21-28
  Determine postoperative speech and swallowing using the Performance Status Scale for Head and Neck (PSS-HN)
Oral Diet | Once each at the following timepoints: 1-2 week preoperatively, postoperative day 7-10, postoperative day 21-28
  Determine food consistencies achieved at short post-operative follow up (per PSS-HN)
Feeding Tube Placement | 30 days postoperatively
  Determine rate of feeding tube placement
Blood Glucose | 30 days postoperatively
  Determine blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Yao, MD FRCSC, Principal Investigator — University Health Network, Toronto; John R de Almeida, MD MSc FRCSC, Study Director — University Health Network, Toronto; Michael Xie, MD FRCSC, Study Chair — University Health Network, Toronto; Rosemary Martino, Ma MSc PhD, Study Chair — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, randomization, primary and secondary outcomes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: May 2027-May 2037
Access Criteria: IPD can be shared on a case by case basis by contacting the principal investigator, data will be de-identified, extent of data will be determined and decided upon by the principal investigator, data will be shared via secure email and data transfer agreement

REFERENCES:
- [Derived] Xie M, de Almeida J, Goldstein D, Martino R, Liu YF, Allen B, Xu W, Hueniken K, Yao CM. Buccal fat applied to transoral robotic lateral oropharyngectomy defects to lessen radical tonsillectomy pain (BOLT): a single-centre, phase II, parallel, randomised control trial study protocol. BMJ Open. 2025 Dec 12;15(12):e106125. doi: 10.1136/bmjopen-2025-106125. PMID 41387003